CLINICAL TRIAL: NCT07358013
Title: Isolation and Characterization of Endothelial Colony Forming Cells (ECFCs) in Patients Diagnosed With Von Willebrand Disease, Acquired Von Willebrand Syndrome and Healthy Subjects
Brief Title: Endothelial Colony-Forming Cells in Patients With VWD, AVWS and Healthy Subjects
Acronym: ECFCs/2022
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 3387 n.6569
Record Dates: First submitted 2025-12-17; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Von Willebrand Disease (VWD); Acquired Von Willebrand Disease
Keywords: von Willebrand disease; von Willebrand factor; ex vivo; endothelial colony forming cells (ECFCs)
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Plasma samples for VWF testing (all enrolled subjects).
  * Peripheral blood-derived ECFCs, cryopreserved after successful isolation (all enrolled subjects).
  * Blood sample for VWF genetic analysis (patients without prior molecular characterization).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- von willebrand disease/ Acquired von Willebrand disease patients: Patients with a confirmed diagnosis of VWD or AVWS. Participants will undergo peripheral blood sample collection for plasma VWF measurements and ECFCs isolation and characterization. In patients with VWD without prior molecular characterization, an additional blood sample will be collected for genetic analysis.
  Interventions: Diagnostic Test: Blood sample collection for VWF measurements in plasma; Other: Blood sample collection for ECFC isolation and characterization; Other: Genetic testing of VWF
- Healthy donors: Healthy volunteers with no personal or family history of bleeding or thrombotic disorders, serving as the reference population for the study. Participants will undergo peripheral blood sample collection plasma VWF measurements and ECFCs isolation and characterization.
  Interventions: Diagnostic Test: Blood sample collection for VWF measurements in plasma; Other: Blood sample collection for ECFC isolation and characterization

INTERVENTIONS:
Diagnostic Test: Blood sample collection for VWF measurements in plasma — Plasma samples will be collected for the measurement of VWF levels.
Other: Blood sample collection for ECFC isolation and characterization — Blood samples will be collected to isolate ECFCs and perform their subsequent characterization.
Other: Genetic testing of VWF — An additional blood sample will be collected for VWF genetic testing in patients with VWD without prior molecular characterization.
  Groups: von willebrand disease/ Acquired von Willebrand disease patients

SUMMARY:
The goal of this observational study is to learn how endothelial colony-forming cells (ECFCs) behave in people with von Willebrand disease (VWD), acquired von Willebrand syndrome (AVWS), and in healthy individuals.

DETAILED DESCRIPTION:
The study aims to establish a reference population of endothelial colony-forming cells (ECFCs) from healthy subjects and compare them with ECFCs derived from patients with VWD/AVWS.

This comparison will help identify cellular and molecular alterations underlying qualitative and quantitative VWF defects. Findings will be correlated with clinical and biochemical data to clarify disease mechanisms.

Study Design: This is a national, monocentric, non-pharmacological study promoted by Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico and coordinated by SC Medicina - Emostasi e Trombosi.

Enrollment: Patients with a prior diagnosis of VWD or AVWS referred to the Angelo Bianchi Bonomi Hemophilia and Thrombosis Center will be contacted for scheduled enrollment. Historical clinical, biochemical, and molecular data will be reviewed, informed consent obtained, and a study-specific blood sample collected to confirm VWF levels and isolate ECFCs.

Healthy volunteers with no history of bleeding or thrombotic disorders will be enrolled in a number equal to that of the patient group. After a brief health interview and informed consent, they will undergo the same blood collection procedures as patients.

Sample collection:

Participants will undergo blood withdrawal for the following procedures:

* Eight milliliters of plasma in sodium citrate will be aliquoted and stored at -80 °C. These samples will be used to confirm patients' diagnoses and, for controls, to measure VWF levels.
* Genetic analysis: one citrate tube will be collected for congenital patients without previous molecular characterization.
* A total of 50 ml of blood in lithium heparin will be drawn for ECFC isolation following the previously published protocol. The isolation procedure will be performed within 3 h of sample collection. In case of unsuccessful isolation, participants may be asked to undergo a second and final blood draw.

Plasma sample testing common to all enrolled subjects: all enrolled subjects will undergo standard plasma testing, including VWF antigen, FVIII activity, VWF activity (VWF:RCo or VWF:GPIbR), VWF collagen-binding activity, and VWF propeptide.

Low-resolution VWF multimer analysis will be performed using either the in-house method or a the semi-automated system.

Procedure to be Performed on ECFCs (common to all enrolled subjects):

* ECFC isolation will follow a modified version of the protocol by Martin-Ramirez et al. (Nat Protoc. 2012;7:1709-1715).
* Flow cytometry will be performed to confirm endothelial lineage.
* Confocal immunofluorescence microscopy will be performed by plating ECFCs on rat tail collagen type I-coated glass slides. Selected markers will include DAPI for nuclei, VWF, and other endothelial markers.
* Basal and stimulated VWF secretion (after histamine or PMA exposure) will be assessed by measuring VWF:Ag levels in culture media and cell lysates using an in-house ELISA.
* VWF multimeric analysis will be performed using the same procedure applied to plasma samples.
* RNA expression analysis will include RNA isolation, first-strand cDNA synthesis, and quantitative real-time PCR for VWF and additional markers using pre-designed TaqMan® assays (ThermoFisher Scientific), normalized to GAPDH or other housekeeping genes.

Assay limited to ECFCs isolated from group B patients and selected controls:

Angiogenesis assay will be performed using Matrigel (Corning). ECFCs obtained from healthy volunteers will be used to establish the assay conditions and will serve as a reference for the analysis of ECFCs isolated from patients.

Assay limited to ECFCs isolated form group C and selected controls: sub-group study:

Inhibition of the mutant allele using small interfering RNA (siRNA) will be performed in a patient selected based on the specific genetic defect (type 2A mutation). ECFCs from this patient will be transfected with a customized siRNA targeting the mutant allele, while a commercial VWF-specific siRNA and a negative control siRNA will be used as controls on both type 2A ECFCs and healthy volunteer-derived ECFCs. All ECFC procedures will be repeated after siRNA silencing, and results will be compared with those obtained from healthy control ECFCs.

Data analysis Continuous variables will be reported as median and interquartile range, whereas categorical variables will be presented as counts and percentages. Laboratory results will be expressed as mean and standard deviation. Comparisons will be performed using one-way ANOVA or Kruskal-Wallis tests, depending on whether variables follow a normal or non-normal distribution. A p-value <0.05 will be considered statistically significant.

Correlation analyses between VWF mRNA expression levels and VWF secreted in cell media, cell lysates, and corresponding plasma VWF levels will be conducted using Pearson's or Spearman's rank correlation, as appropriate.

When available, analyses will be performed using more than one ECFC clone from each enrolled subject.

ELIGIBILITY:
Inclusion Criteria for patients:

Patients with von Willebrand disease (VWD) or acquired von Willebrand syndrome (AVWS)

Age ≥ 16 years.

Previous diagnosis of von Willebrand disease or acquired von Willebrand syndrome, defined as one of the following:

Group A - Type 1 VWD:

VWF levels ≤ 30 IU/dL, regardless of bleeding history, or

VWF levels ≤ 0.50 IU/mL in the presence of abnormal bleeding.

Group B - Congenital or acquired VWD (VWD or AVWS):

Diagnosis of congenital or acquired VWD, with or without gastrointestinal bleeding.

Group C - Subgroup study (Type 2A VWD):

One patient with type 2A VWD selected for a dedicated sub-study involving allele-specific siRNA silencing of the mutant allele.

Ability and willingness to provide written informed consent.

For patients without prior molecular characterization: willingness to undergo VWF gene sequencing and to sign the related informed consent.

Inclusion criteria for healthy volunteers

* No prior diagnosis of VWD, bleeding disorders, or thrombotic disorders.
* Willingness to donate blood for study procedures.
* Ability and willingness to provide written informed consent.
* Age ≥ 18 years.

Exclusion criteria for both patients and healthy volunteers:

* Pregnancy.
* Anemia, as determined at screening or based on medical history.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include the enrollment of subjects with a previous diagnosis of VWD or AVWS and a group of healthy volunteers (controls). Patients will be selected among those referred at Angelo Bianchi Bonomi Haemophilia and Thrombosis Center, with a previous diagnosis of VWD or AVWS.
  Healthy volunteers, defined as individuals without a previous diagnosis of bleeding or thrombotic disorders will be enrolled in equal number to cases with the aim of creating a ECFCs reference group. At enrollment, controls will undergo an interview to confirm their health status, they will be asked to sign the informed consent and then they will undergo a blood withdrawal necessary to confirm plasma VWF levels and to isolate ECFCs as already described for patients.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
ECFCs isolation and characterization | 42 weeks from enrollment start
  Assessment of differences between ECFCs derived from patients with VWD or AVWS and healthy controls.
  Basal and stimulated VWF production and secretion by ECFCs, including basal VWF levels in culture media and cell lysates and stimulated VWF release following exposure to biological or chemical compounds, measured by ELISA (IU/dL) and compared between patients with VWD/AVWS and healthy controls.
  VWF mRNA expression levels in ECFCs, assessed by quantitative real-time PCR and expressed as ΔΔCt, compared between patients with VWD/AVWS and healthy controls.

SECONDARY OUTCOMES:
Correlation of ECFC VWF Antigen Protein and mRNA Levels with Plasma and Platelet VWF Antigen/Activity Levels and Molecular Defect. | 42 weeks from enrollment start
  Correlation analyses between ECFC-derived VWF parameters and circulating VWF levels in corresponding patients with VWD, AVWS, and healthy controls. ECFC-derived VWF antigen levels in culture media and cell lysates (IU/dL), measured by ELISA, and VWF mRNA expression levels in ECFCs (ΔΔCt), assessed by quantitative real-time PCR, will be correlated with plasma and platelet VWF antigen and activity levels (IU/dL). All ECFC-derived and circulating VWF parameters will additionally be analyzed in relation to the specific underlying molecular defect.
Comparison of angiogenic properties of ECFCs from patients with VWD/AVWS and healthy controls | 42 weeks from enrollment start
  Angiogenic properties of ECFCs will be assessed using an in vitro Matrigel tube formation assay and compared between patients with type 2 or type 3 VWD or AVWS and healthy controls. Quantitative parameters will include total tube length (μm), number of tubes, number of branches, and number of meshes.
Evaluation of Allele-Specific siRNA to Restore Normal VWF Levels in Type 2A VWD | 42 weeks from enrollment start
  Allele-specific small interfering RNA (siRNA) will be evaluated in endothelial ECFCs derived from a patient with type 2A VWD to assess whether selective inhibition of the mutant allele restores normal VWF expression and secretion. All analyses will be performed before and after siRNA transfection. The following parameters will be assessed: VWF mRNA expression levels, assessed by quantitative real-time PCR and expressed as ΔΔCt (relative expression); VWF protein levels in ECFC culture media, measured by ELISA (IU/mL).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, A.B.Bonomi Hemophilia and Thrombosis Center, Milan, Italy

IPD SHARING:
Plan to Share IPD: No